CLINICAL TRIAL: NCT03630133
Title: A Prospective, Open-Label, Single-Arm, Single-Center Study of Intraosseous Basivertebral Nerve Ablation for the Treatment of Chronic Low Back Pain
Brief Title: Intraosseous Basivertebral Nerve Ablation for the Treatment of Chronic Low Back Pain
Acronym: CLBP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Combined with NCT03266107
Sponsor: Relievant Medsystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP 0008
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intracept System Ablation (Experimental): Single Arm
  Interventions: Device: Intracept System Ablation

INTERVENTIONS:
Device: Intracept System Ablation — Radiofrequency ablation using Intracept System

SUMMARY:
Objective of study is to evaluate the procedural success rate, clinical effectiveness, and heath-economic profile using the Intercept Intraosseous Nerve Ablation System in adult subjects with chronic low back pain in the post-market setting

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm, single-center study. There is no randomization or blinding. Subjects will receive the Intercept System procedure to treat one or two motion segments at L3/L4, L4/L5, or L5/S1 as identified by Modic Type 1 or 2 changes.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature subjects age 25-70 years, inclusive
* Chronic lower back pain for at least six months
* Failure to respond to at least six months of non-operative conservative management
* Oswestry Disability Index (ODI) at time of evaluation of at least 30 points
* Modic changes (Type 1 or 2) in at least one vertebral endplate, at one or more levels from L3 to S1

Exclusion Criteria:

* Radicular pain by history or evidence of pain neurological deficit within the past one year.
* Previous surgery performed on the lumbar spine
* Current or history of symptomatic spinal stenosis
* Current or history of osteoporotic or tumor-related vertebral body compression fracture
* Current or history of vertebral cancer or spinal metastasis
* Current or history of spinal infection
* Metabolic bone disease
* BMI greater or equal to 40
* Any radiographic evidence of other important back pathology
* MRI evidence of Modic changes, Type 1 or 2 at greater than 3 vertebral bodies or at non-consecutive levels, or at vertebral bodies other than L3 to S1
* Any back pathology related to trauma, evidence of vertebral compression fracture or other spinal pathology that could affect assessment of response to back pain
* Subjects who are bed bound
* Demonstrates 3 or more Waddell's signs of Inorganic Behavior
* Any evidence of current systemic infection

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 3 months
  Mean change in Oswestry Disability Index Score from baseline to 3 months post-treatment. Scale is measured from 0 to 100, better to worse respectively.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 3, 6, 9, and 12 months
  Mean change in Visual Analog Scale (VAS) pain score from baseline to 3, 6, 9 and 12 months post-treatment. Scale is measured from 0 to 10, better to worse respectively.
Oswestry Disability Index (ODI) | 6, 9, and 12 months
  Mean change in Oswestry Disability Index (ODI) score from baseline to 6, 9 and 12 months post-treatment. Scale is measured from 0 to 100, better to worse respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Macadaeg, MD, Principal Investigator — Indiana Spine Group
Locations (1):
- Indiana Spine Group, Carmel, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: At the completion of trial
URL: http://clbpstudy.com